CLINICAL TRIAL: NCT04803461
Title: Catecholamines Level in Urine and Serum in Stable Non-segmental Vitiligo Patients Before and After Excimer Light
Brief Title: Catecholamines Level in Vitiligo Patients Before and After Excimer Light
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Marwa sayed ali, principle investigator, Assiut University
Other Study IDs: CLIVP
Record Dates: First submitted 2021-03-13; First posted 2021-03-17 (Actual); Last update posted 2021-03-17 (Actual); Status verified 2021-03

CONDITIONS: Vitiligo, Generalized
MeSH Terms: conditions — Vitiligo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine Serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum and urinary catecholamines — estimation of level of serum and urinary catecholamines before and after excimer light treatment for patient with non segmental vitiligo.

SUMMARY:
Vitiligo is an acquired cutaneous disorder of pigmentation, with a 1-2% incidence worldwide, without predilection for sex or race. People affected by vitiligo have a vast reduction of quality of life, caused by the color contrast between healthy pigmented skin and the depigmented vitiligo patches due to death of melanocytes, which may cause psychological problems to the patient.

DETAILED DESCRIPTION:
Despite much research, the etiology of vitiligo and the causes of melanocyte death are not clear. Conventionally, there have been three hypotheses to explain the pathogenesis of vitiligo: neural, immune and self-destructive, but none can completely explain the disease and are probably interrelated.

From therapeutic and prognostic viewpoint, vitiligo is broadly classified in two major subtypes, segmental vitiligo (SV) including focal lesions confined to a segment of the body that does not progress towards generalized disease; and non-segmental vitiligo (NSV) which comprises all generalized usually symmetrical forms, including acrofacial vitiligo.

The increased release of catecholamines (CA) from the autonomic nerve endings in the micro-environment of melanocytes in the affected skin areas might be involved in the aetiopathogenesis of vitiligo through two main mechanisms: a direct cytotoxic action of CA and/or their o-diphenol catabolites and an indirect action, skin and mucosa arterioles possess receptors, activation of which by CA discharge may cause a severe vasoconstriction, leading to epidermal and dermal hypoxia with excessive production of toxic oxyradicals generated by different pathways.In both cases, a genetic predisposition due to insufficient radical scavengers in the affected areas should be taken into account.

First line of non-surgical therapy includes topical corticosteroid therapy and phototherapy (solar exposition, Psoralen + UVA (PUVA), narrowband UVB (NB-UVB). (8-10). The NB-UVB is now considered as the best treatment for extensive vitiligo vulgaris due to its relatively good efficacy and excellent tolerance .

Contrary to the majority of laser devices, the 308-nm excimer laser is not a ''destructive'' form of therapy but induces photobiological effects similar to selective UVB phototherapy (311-312 nm).As for UVB phototherapy, it could be judged that the efficiency of the 308-nm excimer laser in treating vitiligo depends on immunomodulatory effects (induction of the secretion of cytokines, T-lymphocytes apoptosis) and stimulation of melanocyte migration and proliferation from the niche located in hair follicles. The 308-nm excimer laser allows a selective treatment of the lesions. This device has already shown interesting results in post-resurfacing leukoderma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with clinically stable non-segmental vitiligo of different ages and sex treated with excimer light

Exclusion Criteria:

* Pregnant and lactating women.

  * Personal history of hypertrophic scarring, melanoma or other skin cancer.
  * Immunosuppression or taking immunosuppressive or photosensitizing drugs, and phototherapy or any other vitiligo treatment during the last 3 months.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Our study will include 21 stable non segmental vitiligo patients subjected to excimer light treatment .All patients will be recruited from the outpatient clinic of dermatology and andrology department of Assiut University.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-09-30 (Estimated)

PRIMARY OUTCOMES:
serum and urinary catecholamine level in stable non segmental vitiligo patients | three months
  Lesions will be Patients will be treated by Excimer light twice weekly for a maximum of 20 sessions
  * Catecholamines level will be measured in urine and serum before beginning of sessions.
  * catecholamines level in urine and serum will be measured after completion of sessions.

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Kent G, Al'Abadie M. Psychologic effects of vitiligo: a critical incident analysis. J Am Acad Dermatol. 1996 Dec;35(6):895-8. doi: 10.1016/s0190-9622(96)90112-7. PMID 8959947
- [Background] Parsad D, Pandhi R, Dogra S, Kanwar AJ, Kumar B. Dermatology Life Quality Index score in vitiligo and its impact on the treatment outcome. Br J Dermatol. 2003 Feb;148(2):373-4. doi: 10.1046/j.1365-2133.2003.05097_9.x. No abstract available. PMID 12588405
- [Background] Westerhof W, d'Ischia M. Vitiligo puzzle: the pieces fall in place. Pigment Cell Res. 2007 Oct;20(5):345-59. doi: 10.1111/j.1600-0749.2007.00399.x. PMID 17850508
- [Background] Gauthier Y, Cario Andre M, Taieb A. A critical appraisal of vitiligo etiologic theories. Is melanocyte loss a melanocytorrhagy? Pigment Cell Res. 2003 Aug;16(4):322-32. doi: 10.1034/j.1600-0749.2003.00070.x. PMID 12859615
- [Background] Morrone A, Picardo M, de Luca C, Terminali O, Passi S, Ippolito F. Catecholamines and vitiligo. Pigment Cell Res. 1992 Mar;5(2):65-9. doi: 10.1111/j.1600-0749.1992.tb00003.x. PMID 1321419
- [Background] Cucchi ML, Frattini P, Santagostino G, Orecchia G. Higher plasma catecholamine and metabolite levels in the early phase of nonsegmental vitiligo. Pigment Cell Res. 2000 Feb;13(1):28-32. doi: 10.1034/j.1600-0749.2000.130106.x. PMID 10761993
- [Background] Mofty ME, Zaher H, Esmat S, Youssef R, Shahin Z, Bassioni D, Enani GE. PUVA and PUVB in vitiligo--are they equally effective? Photodermatol Photoimmunol Photomed. 2001 Aug;17(4):159-63. doi: 10.1034/j.1600-0781.2001.170403.x. PMID 11499536
- [Background] Scherschun L, Kim JJ, Lim HW. Narrow-band ultraviolet B is a useful and well-tolerated treatment for vitiligo. J Am Acad Dermatol. 2001 Jun;44(6):999-1003. doi: 10.1067/mjd.2001.114752. PMID 11369913
- [Background] Taneja A. Treatment of vitiligo. J Dermatolog Treat. 2002 Mar;13(1):19-25. doi: 10.1080/09546630252775207. PMID 12006134
- [Background] Friedman PM, Geronemus RG. Use of the 308-nm excimer laser for postresurfacing leukoderma. Arch Dermatol. 2001 Jun;137(6):824-5. No abstract available. PMID 11405786
- [Background] Ostovari N, Passeron T, Zakaria W, Fontas E, Larouy JC, Blot JF, Lacour JP, Ortonne JP. Treatment of vitiligo by 308-nm excimer laser: an evaluation of variables affecting treatment response. Lasers Surg Med. 2004;35(2):152-6. doi: 10.1002/lsm.20057. PMID 15334620
- [Background] Lilly E, Lu PD, Borovicka JH, Victorson D, Kwasny MJ, West DP, Kundu RV. Development and validation of a vitiligo-specific quality-of-life instrument (VitiQoL). J Am Acad Dermatol. 2013 Jul;69(1):e11-8. doi: 10.1016/j.jaad.2012.01.038. Epub 2012 Feb 25. PMID 22365883
- [Background] Rossiter ND, Chapman P, Haywood IA. How big is a hand? Burns. 1996 May;22(3):230-1. doi: 10.1016/0305-4179(95)00118-2. PMID 8726264
- [Background] Schallreuter KU, Wood JM, Lemke KR, Levenig C. Treatment of vitiligo with a topical application of pseudocatalase and calcium in combination with short-term UVB exposure: a case study on 33 patients. Dermatology. 1995;190(3):223-9. doi: 10.1159/000246690. PMID 7599386